CLINICAL TRIAL: NCT05354271
Title: Impact of High-intensity Interval Training in Patients With Atrial Fibrillation: Understanding of the Underlying Cardiovascular Mechanisms
Brief Title: High-intensity Interval Training in Patients With Atrial Fibrillation
Acronym: HIIT-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Liverpool Centre for Cardiovascular Science (Unknown); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21LJMUSPONSOR060
Record Dates: First submitted 2021-12-02; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-11

CONDITIONS: Atrial Fibrillation
Keywords: Exercise training; High-intensity interval training; Cardiovascular function; Atrial fibrillation burden; Secondary prevention; Aerobic training
MeSH Terms: conditions — Atrial Fibrillation | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training (Experimental): Patients will cycle or walk/run four intervals of four-min at high intensity with the aim to reach 80-90% of peak oxygen consumption, 90-95% of peak heart rate, 15-17 Borg scale, shortness of breath). Each interval is separated by a three-min active recovery, at 50-60% of peak oxygen consumption or 70-75% of peak heart rate. Total exercise time will be 38 min including the warm-up and cool-down.
  Interventions: Other: High-intensity interval training
- Moderate-intensity continuous training (Active Comparator): Patients will cycle or walk/run continuously at moderate intensity (50-60% of peak oxygen consumption, 70-75% of peak heart rate) for 37 min. Total exercise time will be 47 min for the moderate-intensity continuous training group including warm-up and cool-down (isoenergetic compared to high-intensity interval training).
  Interventions: Other: Moderate-intensity continuous training
- Control (No Intervention): The control group will continue their habits without increasing the level of physical activity nor participate to any supervised exercise training.

INTERVENTIONS:
Other: High-intensity interval training — Patients will cycle or walk/run four intervals of four-min at high intensity with the aim to reach 80-90% of peak oxygen consumption, 90-95% of peak heart rate, 15-17 Borg scale, shortness of breath). Each interval is separated by a three-min active recovery, at 50-60% of peak oxygen consumption or 70-75% of peak heart rate. Total exercise time will be 38 min including the warm-up and cool-down.
  Arms: High-intensity interval training
Other: Moderate-intensity continuous training — Patients will cycle or walk/run continuously at moderate intensity (50-60% of peak oxygen consumption, 70-75% of peak heart rate) for 37 min. Total exercise time will be 47 min for the Moderate-intensity continuous training group including warm-up and cool-down (isoenergetic compared to high-intensity interval training).
  Arms: Moderate-intensity continuous training

SUMMARY:
A key characteristic of the heart is its regular rhythm. When the heart is exposed to irregular electric impulses, such as with atrial fibrillation (AF), detrimental effects can occur affecting the ability of the heart to pump blood. AF affects more than 33 million individuals worldwide, and places individuals at increased risk for stroke, heart failure and death. Of note, being fit seems to protect the long-term severity of AF, and individuals with AF who improved their aerobic fitness seem to decrease their severity of atrial fibrillation. Although exercise training is known to improve aerobic fitness, there are limited data investigating the benefits of an exercise training program on the reduction of AF burden.

Once AF is present, regular exercise in these patients reduces the risk for developing cardiovascular events. Moreover, exercise training at high-intensity seems to bring greater adaptations in cardiac patients. This effect may be related to improvements in cardiovascular function and structure. No previous study has explored this possibility in patients with AF. Therefore, I will assess cardiac function and blood vessel quality before and after exercise training (at high- and moderate-intensities) in patients with AF. Better insight into how intensity of exercise training could affect the heart and the blood vessels can lead to better exercise recommendations in this population.

This project will contribute to improved clinical care for patients with AF, specifically related to the prescription of the optimal dose and type of exercise. This may result in fewer complications, improved quality of life, and lower socio-economic/healthcare costs.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common clinically significant arrhythmia, affecting more than 33 million individuals worldwide. AF leads to structural and electrical remodeling in both the atria and ventricles and is strongly related to an increased risk of stroke, heart failure and death. The CARDIO-FIT study demonstrated that AF patients with a higher baseline aerobic fitness were almost 3 times more likely to maintain arrhythmia freedom after a 4-year follow-up; also, AF patients who gained more than 2 metabolic equivalents (METs, aerobic fitness) were more than two-fold more likely to maintain sinus rhythm.

High-intensity exercise training and atrial fibrillation. Each METs gained was associated with a 9% decline in the risk of arrhythmia recurrence. From studies performed in patients with cardiovascular disease, high-intensity interval training (HIIT) seems to bring at least similar or greater improvements in aerobic fitness compared to a moderate-intensity continuous training (MICT). Moreover, in patients with AF, time in AF was reduced of -3.3±7.2% after 12 weeks of HIIT compared to an increased time in AF of 4.2±11.8% in a control group without exercise. Whilst this highlights the potency of HIIT, no previous study has directly compared the effects of HIIT vs. MICT in AF patients on AF burden.

Cardiovascular physiological mechanism(s). Patients with AF exhibit cardiac and vascular dysfunction. However, exercise training improves cardiac and vascular function in human, but the effects are unknown in AF patients. This knowledge is important to improve management of patients with AF with an optimal training prescription. Research on long-term effects and safety related to high-intensity exercise in AF patients is therefore warranted. The findings of the optimal training prescription will help us to update and improve the current guidelines.

Building on the latest scientific insights, the overall aim of this proposal is to determine the optimal intensity for reducing the AF burden. Moreover, the understanding of the underlying mechanisms could help us to determine the cardiovascular adaptations related to exercise training (HIIT or MICT).

Taken together, this study will answer these two questions:

1. What is the best exercise intensity for reducing the time in AF?
2. What are the underlying cardiovascular mechanisms associated with any training related decrease in AF burden? Objectives. Objective 1. High-intensity interval training and AF: The investigators will compare the effects of HIIT and MICT on the burden of AF to test the hypothesis that HIIT decreases the time in AF to a greater extent than MICT.

Objective 2. Cardiovascular physiological mechanisms: The investigators will assess cardiovascular function in all AF patients before and after the training intervention, to test the hypothesis that HIIT is associated with greater cardiovascular adaptation compared to MICT.

Methods. Experimental design: The investigators will perform a 3-arm randomised controlled trial to answer the first research question. The investigators will compare regular care (control group) with regular care + HIIT and regular care + MICT in a total of 60 stable outpatients with non-permanent AF in need for rhythm control (catheter ablation or cardioversion) on the pre-procedure burden of AF, and post-procedure recurrence. When participants are listed on the waiting list for the ablation procedure, they will be assigned to control or HIIT or MICT in a randomized order. The waiting list is approximately 3 months, so patients would have the exercise program for at least 3 months prior to the rhythm control procedure, and continue for 3 months post-procedure to assess AF recurrence. To answer the second research question, the investigators will perform cardiac and vascular functions measurements at baseline, 3 months, and 6 months training intervention in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Presence of non-permanent AF
* > 18 years old

Exclusion Criteria:

* Performing endurance training at high intensity >2 times/week or at moderate intensity >3 times/week;
* Previous cardiac surgery not related to AF;
* LVEF <45%;
* Severe coronary artery disease non-suitable for revascularization;
* Significant cardiac valve disease;
* Implanted cardiac pacemaker;
* And restriction to cardiopulmonary exercise testing or severe intolerance to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-01-27 (Estimated); Study Completion 2023-01-27 (Estimated)

PRIMARY OUTCOMES:
Change in burden of atrial fibrillation | baseline and 3 months post rhythm control procedure
  Burden of atrial fibrillation (number of episodes) continually measured, and reported by the patient. Measured by Huawei Band 4 and 6

SECONDARY OUTCOMES:
Maximal oxygen uptake | baseline and 3 months post rhythm control procedure
  VO2peak
Peripheral endothelial function | baseline and 3 months post rhythm control procedure
  FMD
Carotid structure | baseline and 3 months post rhythm control procedure
  IMT
Central endothelial function | baseline and 3 months post rhythm control procedure
  CAR
Health related quality of life | baseline and 3 months post rhythm control procedure
  Measured with the Medical Outcome Survey Short Form-36 (SF-36) questionnaire
Health related quality of life | baseline and 3 months post rhythm control procedure
  Measured with the Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire
Health related quality of life | baseline and 3 months post rhythm control procedure
  Measured with the modified Mayo AF-Specific Symptom Inventory (mMAFSI) questionnaire
Health related quality of life | baseline and 3 months post rhythm control procedure
  Measured with the HeartQoL questionnaire
Physical activity level | baseline and 3 months post rhythm control procedure
  Steps, sedentary time, light (< 3 METs), moderate (3-<6 METs) and vigorous (≥6 METS) physical activities, measured with the Huawei bands for 14 nights and days (24h)
Resting atrial and ventricular function | baseline and 3 months post rhythm control procedure
  Atrial and ventricular function including left ventricular function, volume, dimension of the cavities, wall thickness, blood and tissue velocities measured by echocardiography
Myocardial strain | baseline and 3 months post rhythm control procedure
  GLS, circumferential and radial strain measured by echocardiography
Strain-area loop | baseline and 3 months post rhythm control procedure
  Relation between changes in volume and strain measured by echocardiography
Atrial and ventricular function during exercise | baseline and 3 months post rhythm control procedure
  Atrial and ventricular function including left ventricular function, volume, dimension of the cavities, wall thickness, blood and tissue velocities measured by echocardiography during exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool Centre for Cardiovascular Sciences, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
It is the first training intervention study in our Lab, so we haven't decided yet and it could be an option if other training studies are conducted.